CLINICAL TRIAL: NCT02408523
Title: A Double-blind, Randomized, Placebo-controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Lacosamide as Adjunctive Therapy for Uncontrolled Primary Generalized Tonic-Clonic Seizures in Subjects With Idiopathic Generalized Epilepsy
Brief Title: A Study to Assess the Safety and Efficacy of Lacosamide Versus Placebo (a Pill Without Active Medication) in Patients With Idiopathic Generalised Epilepsy Who Are Already Taking Anti-epileptic Medications
Acronym: VALOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0982; 2011-003100-21 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; Epilepsy; Children; Primary Generalized Tonic Clonic seizures; Idiopathic Generalized Epilepsy; Adults
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacosamide (Experimental): Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day are allowed. Maximal dose 400 mg/day for adult subjects and pediatric subjects >= 50 kg.
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric subjects < 30 kg.)
  Lasosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric subjects 30 kg to < 50 kg.)
  Interventions: Drug: Lacosamide Tablet; Drug: Lasosamide Oral Solution
- Placebo (Placebo Comparator): Placebo 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day are allowed. Maximal dose 400mg/day for adult subjects and pediatric subjects >= 50kg.
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric subjects < 30kg.)
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric subjects 30kg to < 50kg.)
  Interventions: Other: Placebo Tablet; Other: Placebo Oral Solution

INTERVENTIONS:
Drug: Lacosamide Tablet — * Active Substance: Lacosamide
  * Pharmaceutical Form: Film-coated Tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Other Names: Vimpat
  Arms: Lacosamide
Drug: Lasosamide Oral Solution — * Active Substance: Lacosamide
  * Pharmaceutical Form: Oral Solution
  * Concentration: 10 mg/ml
  * Route of Administration: Oral use
  Other Names: Vimpat
  Arms: Lacosamide
Other: Placebo Tablet — * Active Substance: Placebo
  * Pharmaceutical Form: Film-coated Tablet
  * Concentration: 50 mg
  * Route of Administration: Oral use
  Arms: Placebo
Other: Placebo Oral Solution — * Active Substance: Placebo
  * Pharmaceutical Form: Oral Solution
  * Concentration: 10 mg/ml
  * Route of Administration: Oral use
  Arms: Placebo

SUMMARY:
Evaluating efficacy & safety of lacosamide versus Placebo in a blinded fashion as add-on Therapy for Primary Generalized Tonic-clonic (PGTC) seizures in subject 4 years of age or greater with idiopathic generalized epilepsy currently taking 1 to 3 antiepileptic drugs. Maximum duration of study drug administration is 28 weeks. Eligible subjects may choose to enter the open-label extension study after completion.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a confirmed diagnosis at least 24 weeks prior to Visit 1 and a disease onset prior to 30 years of age, consistent with idiopathic generalized epilepsy (IGE) experiencing primary generalized tonic-clonic (PGTC) seizures (Type IIE) that are classifiable according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (ILAE, 1981)
* Subject has >=3 PGTC seizures during the 16-week Combined Baseline (12-week Historical Baseline plus 4-week Prospective Baseline)
* If a brain magnetic resonance imaging (MRI)/computed tomography (CT) scan has been performed, there must be no evidence of any progressive abnormality or any lesion likely to be associated with partial-onset seizures
* Subject has been maintained on a stable dose regimen of 1 to 2 non-benzodiazepine marketed antiepileptic drugs (AEDs) with no benzodiazepine AEDs OR 1 benzodiazepine marketed AED with 1 to 2 non benzodiazepine marketed AEDs for at least 28 days prior to Visit 1 with or without additional concurrent stable vagus nerve stimulation (VNS)
* Subjects are required to have had an electroencephalogram (EEG) report consistent with idiopathic generalized epilepsy (eg, generalized 3Hz epileptiform discharges and a normal EEG background) confirmed by a Central Reviewer

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to Lacosamide (LCM)
* Subject meets the withdrawal criteria for SP0982 or is experiencing an ongoing serious adverse event (SAE)
* Subject has an active suicidal ideation as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the 'Since Last Visit' version of the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Subject has >=2x upper limit of normal (ULN) of any of the following: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or >ULN total bilirubin (>=1.5xULN total bilirubin if known Gilbert's syndrome). If subject has elevations only in total bilirubin that are >ULN and <1.5xULN, fractionate bilirubin to identify possible undiagnosed Gilbert's syndrome (ie, direct bilirubin <35%)

For randomized subjects with a Baseline result >ULN for ALT, AST, ALP, or total bilirubin, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the electronic case report form (eCRF).

If subject has >ULN ALT, AST, or ALP that does not meet the exclusion limit at screening, repeat the tests, if possible, prior to dosing to ensure there is no further ongoing clinically relevant increase. In case of a clinically relevant increase, inclusion of the subject must be discussed with the Medical Monitor.

Tests that result in ALT, AST, or ALP up to 25% above the exclusion limit may be repeated once for confirmation. This includes re-screening.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (115):
- United States (27):
  - Sp0982 028, Alabaster, Alabama
  - Sp0982 005, Little Rock, Arkansas
  - Sp0982 018, Irvine, California
  - Sp0982 008, Santa Monica, California
  - Sp0982 031, Colorado Springs, Colorado
  - Sp0982 035, Denver, Colorado
  - Sp0982 036, Danbury, Connecticut
  - Sp0982 011, Jacksonville, Florida
  - Sp0982 013, Panama City, Florida
  - Sp0982 002, Port Charlotte, Florida
  - Sp0982 042, Wellington, Florida
  - Sp0982 015, Boise, Idaho
  - Sp0982 021, Peoria, Illinois
  - Sp0982 045, Springfield, Illinois
  - Sp0982 009, New Orleans, Louisiana
  - Sp0982 007, Bethesda, Maryland
  - Sp0982 010, Waldorf, Maryland
  - Sp0982 025, Golden Valley, Minnesota
  - Sp0982 029, St Louis, Missouri
  - Sp0982 043, New York, New York
  - Sp0982 053, Austin, Texas
  - Sp0982 050, Greenville, Texas
  - Sp0982 034, Houston, Texas
  - Sp0982 047, San Antonio, Texas
  - Sp0982 038, San Antonio, Texas
  - Sp0982 027, Renton, Washington
  - Sp0982 023, Madison, Wisconsin
- Australia (4):
  - Sp0982 981, Parkville, Victoria
  - Sp0982 980, Chatswood
  - Sp0982 985, Heidelberg
  - Sp0982 986, Parkville
- Belgium (3):
  - Sp0982 201, Brussels
  - Sp0982 202, Ghent
  - Sp0982 200, Leuven
- Brazil (7):
  - Sp0982 181, Curitiba
  - Sp0982 180, Florianópolis
  - Sp0982 186, Passo Fundo
  - Sp0982 185, Porto Alegre
  - Sp0982 188, Rio de Janeiro
  - Sp0982 183, São Paulo
  - Sp0982 184, São Paulo
- Bulgaria (2):
  - Sp0982 500, Blagoevgrad
  - Sp0982 501, Sofia
- China (6):
  - Sp0982 971, Beijing
  - Sp0982 976, Changchun
  - Sp0982 975, Chongqing
  - Sp0982 097, Fuzhou
  - Sp0982 973, Hangzhou
  - Sp0982 972, Shanghai
- Czechia (4):
  - Sp0982 550, Ostrava Poruba
  - Sp0982 553, Prague
  - Sp0982 556, Prague
  - Sp0982 552, Zlín
- France (4):
  - Sp0982 255, Bron
  - Sp0982 252, Lille
  - Sp0982 251, Nancy
  - Sp0982 250, Rennes
- Germany (5):
  - Sp0982 305, Berlin
  - Sp0982 303, Erlangen
  - Sp0982 314, Freiburg im Breisgau
  - Sp0982 311, Marburg
  - Sp0982 302, München
- Hungary (2):
  - Sp0982 600, Budapest
  - Sp0982 603, Szeged
- Israel (2):
  - Sp0982 850, Rehovot
  - Sp0982 851, Tel Litwinsky
- Sp0982 351, Torino, Italy
- Japan (14):
  - Sp0982 907, Asaka
  - Sp0982 906, Fukuoka
  - Sp0982 910, Gifu
  - Sp0982 903, Hamamatsu
  - Sp0982 902, Hiroshima
  - Sp0982 913, Itami
  - Sp0982 912, Kagoshima
  - Sp0982 914, Kodaira
  - Sp0982 909, Kokubunji
  - Sp0982 901, Niigata
  - Sp0982 911, Ōmura
  - Sp0982 900, Sapporo
  - Sp0982 908, Shinjuku-Ku
  - Sp0982 904, Shizuoka
- Sp0982 161, Guadalajara, Mexico
- Poland (10):
  - Sp0982 657, Częstochowa
  - Sp0982 655, Gdansk
  - Sp0982 658, Gdynia
  - Sp0982 652, Gliwice
  - Sp0982 651, Katowice
  - Sp0982 653, Katowice
  - Sp0982 654, Katowice
  - Sp0982 656, Tyniec Mały
  - Sp0982 650, Warsaw
  - Sp0982 659, Warsaw
- Sp0982 451, Lisbon, Portugal
- Romania (3):
  - Sp0982 704, Iași
  - Sp0982 707, Iași
  - Sp0982 700, Timișoara
- Russia (7):
  - Sp0982 750, Kazan'
  - Sp0982 758, Pyatigorsk
  - Sp0982 755, Saint Petersburg
  - Sp0982 756, Saint Petersburg
  - Sp0982 752, Samara
  - Sp0982 753, Smolensk
  - Sp0982 757, Yekaterinburg
- Slovakia (2):
  - Sp0982 821, Bardejov
  - Sp0982 823, Hlohovec
- South Korea (3):
  - Sp0982 940, Daegu
  - Sp0982 941, Seoul
  - Sp0982 944, Seoul
- Spain (5):
  - Sp0982 402, Barcelona
  - Sp0982 406, Córdoba
  - Sp0982 407, Madrid
  - Sp0982 404, Málaga
  - Sp0982 403, Seville
- Taiwan (2):
  - Sp0982 961, Taichung
  - Sp0982 960, Taipei

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in April 2015 and concluded in May 2019.
Pre-assignment Details: Completed study was defined as meeting any exit criteria or completing the 24-week Treatment Period with < 2 PGTCS. After Treatment Period participants enrolled either in a 4-week Transition Period (entered EP0012) or up to a 4-week Taper Period and a 30-day Safety Follow-up Period (did not enter EP0012).
  Participant Flow refers to the Safety Set.
Groups:
- Placebo: Placebo 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400 mg/day for adult and pediatric participants >= 50 kg.
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants < 30 kg).
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
- Lacosamide: Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400 mg/day for adult and pediatric participants with more or equal than (>=) 50 kilograms (kg).
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants with less than (<) 30 kg).
  Lasosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
Period: Overall Study
Arm/Group | Placebo | Lacosamide
Started | 121 | 121
Completed Treatment Period | 110 | 103
Enrolled Transition Period | 108 | 101
Enrolled Taper Period | 7 | 9
Enrolled Safety Folllow-up Period | 10 | 11
Completed | 110 | 103
Not Completed | 11 | 18
Not completed — Adverse Event | 4 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Sponsor request | 1 | 0
Not completed — Did not satisfy extension conditions | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which was a subset of the Randomized Set (RS) and consisted of all study participants who had been treated with at least 1 dose of study medication, either LCM or Placebo.
Arm/Group | Placebo | Lacosamide | Total Title
Number analyzed (Participants) | 121 | 121 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 28 | 55
  Between 18 and 65 years | 93 | 92 | 185
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.64 (12.45) | 27.82 (13.13) | 27.73 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 66 | 142
  Male | 45 | 55 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 1 | 2
  Asian | 25 | 18 | 43
  Black | 2 | 2 | 4
  White | 89 | 97 | 186
  Other/Mixed | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to the Second Primary Generalized Tonic Clonic (PGTC) Seizure During the 24-week Treatment Period From Visit 2 (Week 0) to Visit 10 (Week 24)
Description: The primary efficacy variable was the time to the second primary generalized tonic clonic seizure (PGTCS) during the 24-week Treatment Period. Relative difference between groups (Lacosamide vs Placebo) was expressed as Hazard Ratio.
  The indicated measured values are the observed number of events of second PGTCS in the treatment period which form the basis of the statistical analysis of the time to event analysis.
  The hazard ratio compares 2 treatment groups for the times to a specified number of events (125) for the combined treatment groups, and so both the number of events and the times until those events pertain to the computation of the hazard ratio.
  A Hazard Ratio below 1 indicates time to second PGTCS was improved for LCM compared to Placebo.
Time Frame: During the Treatment Period from Visit 2 (Week 0) to Visit 10 (Week 24)
Population: The Full Analysis Set (FAS) was a subset of the Safety Set (SS) that consisted of all study participants with at least 1 seizure diary assessment during the Treatment Period.
  1 patient from the Lacosamide (FAS) group was randomized after the 125th event and did not appear in this analysis.
Measure: Number; unit: events
Groups:
- Placebo (FAS): Placebo 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400mg/day for adult and pediatric participants >= 50 kg.
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants < 30 kg).
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the Full Analysis Set (FAS).
- Lacosamide (FAS): Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400 mg/day for adult and pediatric participants with more or equal than (>=) 50 kilograms (kg).
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants with less than (<) 30 kg).
  Lasosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the FAS.
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 121 | 118
events | 76 | 49
Statistical Analysis 1: Comparison: Placebo (FAS) vs Lacosamide (FAS); Comparison of LCM versus Placebo was based on a Cox proportional hazards regression model with an effect for treatment, stratifying for the following combinations of study participants' Baseline PGTCS frequency and Development from interactive response technology (IRT) (<= 2 per 28 days in the Combined Baseline Period and Pediatric, <= 2 per 28 days in the Combined Baseline Period and Adult, and > 2 per 28 days in the Combined Baseline Period). The reference group was Placebo; Test type: Superiority; p < 0.001, Regression, Cox — Wald's method was used to calculate the p-value, Hazard Ratio (HR) and confidence intervals (CIs); Hazard Ratio (HR) = 0.540, 95% CI 2-sided [0.377 to 0.774]

2. Secondary Outcome: Percentage of Participants With Seizure Freedom for Primary Generalized Tonic Clonic (PGTC) Seizures During the 24-week Treatment Period From Visit 2 (Week 0) to Visit 10 (Week 24)
Description: A seizure-free day from primary generalized tonic clonic seizures (PGTCS) was defined as a day where no PGTCS were reported in the seizure diary and PGTCS were assessed, which was estimated using Kaplan-Meier (KM) methods.
Time Frame: During the Treatment Period from Visit 2 (Week 0) to Visit 10 (Week 24)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 121 | 118
percentage of participants | 17.3 [10.3 to 24.3] | 31.0 [22.4 to 39.6]
Statistical Analysis 1: Comparison: Placebo (FAS) vs Lacosamide (FAS); The key secondary efficacy variable was evaluated using an extended Mantel-Haenszel testing procedure. Baseline PGTCS Frequency from Combined Baseline and development (age from interactive response technology (IRT)) were calculated from IRT; Test type: Superiority; p = 0.011, Mantel Haenszel — Superiority of LCM vs Placebo p-value was based on a chi-square test on 1 degree of freedom; KM seizure free of LCM vs Placebo = 14.1, 95% CI 2-sided [3.2 to 25.1] — Stratified difference in proportion of subjects who are seizure-free from PGTCS on Lacosamide (FAS) vs Placebo (FAS)

3. Secondary Outcome: Time to the First Primary Generalized Tonic Clonic (PGTC) Seizure During the Treatment Period From Visit 2 (Week 0) to Visit 10 (Week 24)
Description: The secondary efficacy variable was the time to the first primary generalized tonic clonic seizure (PGTCS) during the 24-week Treatment Period. Relative difference between groups (Lacosamide vs Placebo) was expressed as Hazard Ratio.
  The indicated measured values are the observed number of events of first PGTCS in the treatment period which form the basis of the statistical analysis of the time to event analysis.
  The hazard ratio compares 2 treatment groups for the times to the number of events for the combined treatment groups, and so both the number of events and the times until those events pertain to the computation of the hazard ratio.
  A Hazard Ratio below 1 indicates time to second PGTCS was improved for LCM compared to Placebo.
Time Frame: During the Treatment Period from Visit 2 (Week 0) to Visit 10 (Week 24)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 121 | 118
events | 97 | 79
Statistical Analysis 1: Comparison: Placebo (FAS) vs Lacosamide (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.012, Regression, Cox — Wald's method was used to calculate the p-value, Hazard Ratio (HR) and confidence intervals (CIs); Hazard Ratio (HR) = 0.683, 95% CI 2-sided [0.507 to 0.921]

4. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) as Reported Spontaneously by the Subject and/or Caregiver or Observed by the Investigator
Description: An AE was any untoward medical occurrence in a patient or clinical investigation study participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational medicinal product (IMP), whether or not related to the IMP.
Time Frame: From Visit 1 (Week -4) to End of Study Period (up to Week 36)
Population: The Safety Set (SS) was a subset of the Randomized Set (RS) and consisted of all study participants who had been treated with at least 1 dose of study medication, either LCM or Placebo.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Placebo 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400mg/day for adult and pediatric participants >= 50 kg.
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants < 30 kg).
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the Safety Set (SS).
- Lacosamide (SS): Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400 mg/day for adult and pediatric participants with more or equal than (>=) 50 kilograms (kg).
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants with less than (<) 30 kg).
  Lasosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the SS.
Arm/Group | Placebo (SS) | Lacosamide (SS)
Number analyzed (Participants) | 121 | 121
percentage of participants | 81.8 | 82.6

5. Secondary Outcome: Plasma Concentrations of Lacosamide
Description: Lacosamide plasma concentration was expressed in micrograms per milliliter (μg/mL).
  Means and standard deviation (SD) were only calculated if at least 2/3 of the concentrations were quantified at the respective timepoint. Values Below Limit of Quantification (BLQ) were replaced by value of 0 in calculations of means and SDs.
Time Frame: During the Treatment Period from Visit 2 (Week 0) to Visit 10 (Week 24)
Population: The Safety Set (SS) was a subset of the Randomized Set (RS) and consisted of all study participants who had been treated with at least 1 dose of study medication, either LCM or Placebo.
  Data not collected from participants in Placebo (SS) Arm/Group.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo (SS) | Lacosamide (SS)
Number analyzed (Participants) | 0 | 121
ug/mL
  Visit 5, Week 6 (Titration) |  | 8.610961 (3.705438)
  Visit 10, Week 24 (Maintenance) |  | 8.074427 (3.948749)
  Early Termination Visit |  | 8.138085 (4.913627)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week 1 to End of Study Period (up to Week 36).
Description: TEAEs counts are for each study period: Treatment Period, Transition Period for participants who entered EP0012 (NCT02408549) and Taper Period followed by Safety Follow-up Period for participants not entering EP0012.
  AEs reported for PBO participants during the Transition Period occur when they have switched to LCM.
Groups:
- Placebo (SS) Treatment Period: Participants received the following treatment during the Treatment Period (Week 0 to Week 24):
  Placebo 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400mg/day for adult and pediatric participants >= 50 kg.
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants < 30 kg).
  Placebo oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the Safety Set (SS).
- Lacosamide (SS) Treatment Period: Participants received the following treatment during the Treatment Period (Week 0 to Week 24):
  Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 50 mg or 100 mg/day were allowed. Maximal dose 400 mg/day for adult and pediatric participants with more or equal than (>=) 50 kilograms (kg).
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 12 mg/kg/day for pediatric participants with less than (<) 30 kg).
  Lasosamide oral solution 10 mg/ml: starting with 2 mg/kg/day, titrations steps (1 mg/kg/day to 2 mg/kg/day; maximal dose 8 mg/kg/day for pediatric participants 30 kg to < 50 kg).
  Participants formed the SS.
- Placebo (SS) Transition Period: At the end of Visit 10 (Week 24)/ Early Termination (ET), study participants who completed the study may have been eligible to participate in an open-label extension study (EP0012). Study participants who chose to enroll in the open-label extension study proceeded to a blinded 4-week Transition Period.
  Participants randomized to Placebo in the Treatment Period transitioned to double-blind Lacosamide:
  Lacosamide 50 mg tablets: starting with 100 mg/day at Week 1. Weekly increase in steps of 100 mg/day until final dose of 400 mg/day at Week 4 for adult and pediatric participants >= 50 kg.
  Lacosamide oral solution 10 mg/ml: starting with 2 mg/kg/day at Week 1. Weekly increase in steps of 2 mg/kg/day until final dose of 8 mg/kg/day at Week 4 for pediatric participants < 30 kg and 0 kg to < 50 kg.
  Participants formed the SS.
- Lacosamide (SS) Transition Period: At the end of Visit 10 (Week 24)/ Early Termination (ET), study participants who completed the study may have been eligible to participate in an open-label extension study (EP0012). Study participants who chose to enroll in the open-label extension study proceeded to a blinded 4-week Transition Period.
  Participants randomized to Lacosaminde in the Treatment Period continued to receive double-blind Lacosamide:
  Lacosamide 50 mg tablets: minim (min) 300 mg/day to maximum (max) 400 mg/day from Week 1 to Week 3 and final dose of 400 mg/day at Week 4 for adult and pediatric participants >= 50 kg.
  Lacosamide oral solution 10 mg/ml: min 8 mg/kg/day to max 12 mg/kg/day from Week 1 to Week 4 for pediatric participants < 30 kg.
  Lacosamide oral solution 10 mg/ml: min 6 mg/kg/day to max 8 mg/kg/day from Week 1 to Week 3 and final dose of 8 mg/kg/day at Week 4 for pediatric participants 30 kg to < 50 kg.
  Participants formed the SS.
- Placebo (SS) Taper Period: Study participants completing Visit 10 (Week 24) or the ET Visit who chose not to continue in EP0012 must have completed an up to 4 weeks blinded taper followed by the End of Taper Visit.
  Participants randomized to Placebo in the Treatment Period continued to receive Placebo:
  Placebo 50 mg tablets: starting with maximum dose achieved during the Treatment Period. Weekly decrease in steps of 100 mg/day until no treatment received for adult and pediatric participants >= 50 kg.
  Placebo oral solution 10 mg/ml: starting with maximum dose achieved during the Treatment Period. Weekly decrease in steps of 2 mg/kg/day or 3 mg/kg/day until no treatment received for pediatric participants < 30 kg and 0 kg to < 50 kg.
  Participants formed the SS.
- Lacosamide (SS) Taper Period: Study participants completing Visit 10 (Week 24) or the ET Visit who chose not to continue in EP0012 must have completed an up to 4 weeks blinded taper followed by the End of Taper Visit.
  Participants randomized to Lacosamide in the Treatment Period continued to receive Lacosamide:
  Lacosamide 50 mg tablets: starting with maximum dose achieved during the Treatment Period. Weekly decrease in steps of 100 mg/day until no treatment received for adult and pediatric participants >= 50 kg.
  Lacosamide oral solution 10 mg/ml: starting with maximum dose achieved during the Treatment Period. Weekly decrease in steps of 2 mg/kg/day or 3 mg/kg/day until no treatment received for pediatric participants < 30 kg and 0 kg to < 50 kg.
  Participants formed the SS.
- Placebo (SS) Safety Follow-up Period; Lacosamide (SS) Safety Follow-up Period: There was a 30-day (-1/+3 days) Safety Follow-up Period for study participants who completed the End of Taper Visit. The Safety Follow-up Period consisted of a clinic visit 2 weeks after the End of Taper Visit followed 2 weeks later by a telephone contact (TC).
  Participants did not receive any treatment during this period. Participants formed the SS.
Arm/Group | Placebo (SS) Treatment Period | Lacosamide (SS) Treatment Period | Placebo (SS) Transition Period | Lacosamide (SS) Transition Period | Placebo (SS) Taper Period | Lacosamide (SS) Taper Period | Placebo (SS) Safety Follow-up Period | Lacosamide (SS) Safety Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121 | 0/108 | 0/101 | 0/7 | 0/9 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/121 | 8/121 | 0/108 | 3/101 | 0/7 | 0/9 | 1/10 | 1/11
Other Adverse Events (participants affected / at risk) | 41/121 | 60/121 | 27/108 | 5/101 | 3/7 | 2/9 | 0/10 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) Treatment Period (N=121) | Lacosamide (SS) Treatment Period (N=121) | Placebo (SS) Transition Period (N=108) | Lacosamide (SS) Transition Period (N=101) | Placebo (SS) Taper Period (N=7) | Lacosamide (SS) Taper Period (N=9) | Placebo (SS) Safety Follow-up Period (N=10) | Lacosamide (SS) Safety Follow-up Period (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clonic convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) Treatment Period (N=121) | Lacosamide (SS) Treatment Period (N=121) | Placebo (SS) Transition Period (N=108) | Lacosamide (SS) Transition Period (N=101) | Placebo (SS) Taper Period (N=7) | Lacosamide (SS) Taper Period (N=9) | Placebo (SS) Safety Follow-up Period (N=10) | Lacosamide (SS) Safety Follow-up Period (N=11)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 8 (8) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 11 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 7 (10) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 8 (12) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 26 (34) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 17 (17) | 18 (19) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (13) | 16 (18) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02408523/SAP_000.pdf
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT02408523/Prot_001.pdf